CLINICAL TRIAL: NCT03619590
Title: Twinrix [Hepatitis A Inactivated & Hepatitis B (Recombinant) Vaccine] Pregnancy Registry
Brief Title: Twinrix Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201339
Record Dates: First submitted 2018-07-18; First posted 2018-08-08 (Actual); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis
Keywords: Teratogenicity; Pregnancy; Hepatitis B; Twinrix; Prenatal exposure; Hepatitis A
MeSH Terms: conditions — Hepatitis; Teratogenesis; Hepatitis B; Hepatitis A | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Exposure Group: Pregnant women who were exposed to Twinrix within 28 days prior to conception or at any time during pregnancy. Reporting of exposed pregnancies is voluntary and prospective.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — When the pregnancy is reported prospectively, the Registry will collect registration data from the reporter through telephone interview or a short registration form. In the month of the estimated date of delivery, follow-up will be sought by telephone contact or a form mailed to the health professional. Information about maternal events throughout the pregnancy, pregnancy outcome, and neonatal health is requested. Additional follow-up is not sought from subsequent health care providers.

SUMMARY:
The purpose of the Twinrix Pregnancy Registry is to prospectively collect data describing exposure to Twinrix before or during pregnancy, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy.

This is a prospective, voluntary, observational, exposure-registration study. Twinrix is designated as Food and Drug Administration (FDA) Pregnancy Category C, which means that its safety in human pregnancy has not been determined. The Registry is intended to provide an early signal of potential risks in advance of results from formal epidemiologic studies. Registry statistics can supplement animal reproductive toxicology studies and assist clinicians in evaluating the potential risks and benefits of vaccination for individual patients.

DETAILED DESCRIPTION:
The Twinrix Pregnancy Registry will be maintained by GSK Vaccines Clinical Safety and Pharmacovigilance. Enrolment in the Registry will begin at the time of commercial launch of Twinrix in the United States (US). At the time of initiation of the Registry, pre-existing reports of pregnancy from clinical trials will be evaluated and enrolled when the criteria for registration are met. Reporting of exposed pregnancies is voluntary. Pregnancies will be registered following maternal exposure to Twinrix within 28 days prior to conception or during pregnancy. Registration of pregnancies is prospective, i.e., reported during pregnancy before the pregnancy outcome is known. Retrospective reports, in which the pregnancy outcomes are known at the time of reporting, will also be reviewed to assist in the detection of any unusual patterns that may exist among the reported birth defects. However, because there is no denominator from which risk can be calculated, these reports will be excluded from the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Documentation that Twinrix was administered ≤ 28 days before or during pregnancy;
* Confirmation that the pregnancy is being prospectively reported;
* Report made by a patient or a health care professional;
* The timing of the prenatal exposure to Twinrix (no broader than during which trimester);
* A patient identifier that will allow follow-up to be obtained so that the pregnancy outcome can be ascertained;
* Whether the patient was involved in a clinical trial at the time of the exposure;
* Full reporter contact information.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes pregnant women who were exposed to Twinrix within 28 days prior to conception or at any time during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2001-05-18 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population included pregnant women who prospectively reported exposure to Twinrix within 28 days prior to conception or at any time during pregnancy. 245 pregnancies were prospectively registered in the study. 142 pregnancies were lost to follow-up. Outcomes were reported for 103 pregnancies. Hence, the number of subjects started is 103.
Pre-assignment Details: A total of 105 outcomes were reported for 103 pregnancies due to 2 sets of twins, one each from pregnancies with reported exposure during the first trimester and an unspecified trimester, respectively.
Groups:
- Exposure Group: Pregnant women who were exposed to Twinrix within 28 days prior to conception or at any time during pregnancy. Reporting of exposed pregnancies was voluntary and prospective.
Period: Overall Study
Arm/Group | Exposure Group
Started | 103
Completed | 103
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exposure Group
Number analyzed (Participants) | 103
Age, Customized [Count of Participants; unit: Participants]
  ≤ 18 years | 1
  > 18 and < 65 years | 94
  ≥ 65 years | 0
  Age not specified | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Outcomes From Pregnancies With Reported Exposure Within 28 Days of Last Menstrual Period
Description: Participants were followed from registration upon exposure to Twinrix within 28 days prior to conception until data on pregnancy outcome was obtained. Follow-up via telephone or a form mailed to the contact was sought in the month of the estimated date of delivery.
  Pregnancy outcomes were stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration during pregnancy; multiple exposures were classified by the earliest trimester of exposure. Gestational weeks were counted from the date of the last menstrual period. The second trimester was considered to begin at week 14, and the third trimester beginning at week 28.
  Pregnancy outcomes were dichotomized according to the presence or absence of birth defects and further categorized as: Live births, Spontaneous abortions (i.e., pregnancy losses), Induced abortions and Fetal deaths.
Time Frame: From the date of registration until the date of documentation of pregnancy outcome (up to 10 months i.e. 28 days prior to conception till the month of estimated date of delivery)
Population: Analysis was performed on the outcomes reported for the pregnancies with exposure to Twinrix within 28 days prior to conception or at any time during pregnancy. A total of 105 outcomes were reported for 103 pregnancies due to 2 sets of twins, one each from pregnancies with reported exposure during the first trimester and an unspecified trimester.
Measure: Number; unit: Pregnancy Outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 103
Pregnancy Outcomes
  Congenital Abnormalities, Live Birth | 0
  Congenital Abnormalities, Spontaneous Abortion | 0
  Congenital Abnormalities, Fetal Death | 0
  Congenital Abnormalities, Induced Abortion | 0
  No Congenital Abnormalities, Live Birth | 4
  No Congenital Abnormalities, Spontaneous Abortion | 1
  No Congenital Abnormalities, Fetal Death | 1
  No Congenital Abnormalities, Induced Abortion | 0

2. Primary Outcome: Number of Outcomes From Pregnancies With Earliest Reported Exposure During the First Trimester
Description: Participants were followed from registration upon exposure to Twinrix during first trimester of pregnancy until data on pregnancy outcome was obtained. Follow-up via telephone or a form mailed to the contact was sought in the month of the estimated date of delivery.
  Pregnancy outcomes were stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration during pregnancy; multiple exposures were classified by the earliest trimester of exposure. Gestational weeks were counted from the date of the last menstrual period. The second trimester was considered to begin at week 14, and the third trimester beginning at week 28. Pregnancy outcomes were dichotomized according to the presence or absence of birth defects and further categorized as: Live births, Spontaneous abortions (i.e., pregnancy losses), Induced abortions and Fetal deaths.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Pregnancy Outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 103
Pregnancy Outcomes
  Congenital Abnormalities, Live Birth | 3
  Congenital Abnormalities, Spontaneous Abortion | 0
  Congenital Abnormalities, Fetal Death | 0
  Congenital Abnormalities, Induced Abortion | 1
  No Congenital Abnormalities, Live Birth | 60
  No Congenital Abnormalities, Spontaneous Abortion | 7
  No Congenital Abnormalities, Fetal Death | 0
  No Congenital Abnormalities, Induced Abortion | 5

3. Primary Outcome: Number of Outcomes From Pregnancies With Earliest Reported Exposure During the Second Trimester
Description: Participants were followed from registration upon exposure to Twinrix during second trimester of pregnancy until data on pregnancy outcome was obtained. Follow-up via telephone or a form mailed to the contact was sought in the month of the estimated date of delivery.
  Pregnancy outcomes were stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration during pregnancy; multiple exposures were classified by the earliest trimester of exposure. Gestational weeks were counted from the date of the last menstrual period. The second trimester was considered to begin at week 14, and the third trimester beginning at week 28. Pregnancy outcomes were dichotomized according to the presence or absence of birth defects and further categorized as: Live births, Spontaneous abortions (i.e., pregnancy losses), Induced abortions and Fetal deaths.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Pregnancy Outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 103
Pregnancy Outcomes
  Congenital Abnormalities, Live Birth | 2
  Congenital Abnormalities, Spontaneous Abortion | 0
  Congenital Abnormalities, Fetal Death | 0
  Congenital Abnormalities, Induced Abortion | 0
  No Congenital Abnormalities, Live Birth | 11
  No Congenital Abnormalities, Spontaneous Abortion | 0
  No Congenital Abnormalities, Fetal Death | 0
  No Congenital Abnormalities, Induced Abortion | 0

4. Primary Outcome: Number of Outcomes From Pregnancies With Earliest Reported Exposure During the Third Trimester
Description: Participants were followed from registration upon exposure to Twinrix during third trimester of pregnancy until data on pregnancy outcome was obtained. Follow-up via telephone or a form mailed to the contact was sought in the month of the estimated date of delivery.
  Pregnancy outcomes were stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration during pregnancy; multiple exposures were classified by the earliest trimester of exposure. Gestational weeks were counted from the date of the last menstrual period. The second trimester was considered to begin at week 14, and the third trimester beginning at week 28. Pregnancy outcomes were dichotomized according to the presence or absence of birth defects and further categorized as: Live births, Spontaneous abortions (i.e., pregnancy losses), Induced abortions and Fetal deaths.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Pregnancy Outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 103
Pregnancy Outcomes
  Congenital Abnormalities, Live Birth | 0
  Congenital Abnormalities, Spontaneous Abortion | 0
  Congenital Abnormalities, Fetal Death | 0
  Congenital Abnormalities, Induced Abortion | 0
  No Congenital Abnormalities, Live Birth | 1
  No Congenital Abnormalities, Spontaneous Abortion | 0
  No Congenital Abnormalities, Fetal Death | 0
  No Congenital Abnormalities, Induced Abortion | 0

5. Primary Outcome: Number of Outcomes From Pregnancies With Reported Exposure During an Unspecified Trimester
Description: Participants were followed from registration upon exposure to Twinrix during unspecified trimester of pregnancy until data on pregnancy outcome was obtained. Follow-up via telephone or a form mailed to the contact was sought in the month of the estimated date of delivery.
  Pregnancy outcomes were stratified by the trimester of exposure, with an additional stratum for preconception exposure with no subsequent administration during pregnancy; multiple exposures were classified by the earliest trimester of exposure. Gestational weeks were counted from the date of the last menstrual period. The second trimester was considered to begin at week 14, and the third trimester beginning at week 28. Pregnancy outcomes were dichotomized according to the presence or absence of birth defects and further categorized as: Live births, Spontaneous abortions (i.e., pregnancy losses), Induced abortions and Fetal deaths.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Pregnancy Outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 103
Pregnancy Outcomes
  Congenital Abnormalities, Live Birth | 0
  Congenital Abnormalities, Spontaneous Abortion | 0
  Congenital Abnormalities, Fetal Death | 0
  Congenital Abnormalities, Induced Abortion | 0
  No Congenital Abnormalities, Live Birth | 7
  No Congenital Abnormalities, Spontaneous Abortion | 2
  No Congenital Abnormalities, Fetal Death | 0
  No Congenital Abnormalities, Induced Abortion | 0

ADVERSE EVENTS:
Description: No safety data was collected in the study.
Arm/Group | Exposure Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT03619590/Prot_SAP_000.pdf